CLINICAL TRIAL: NCT03439046
Title: A Phase IIIb, Open-label, Local, Multicenter Study of the Molecular Features of Postmenopausal Women With Hormone Receptor-positive (HR+) HER2-negative Advanced Breast Cancer on First-line Treatment With Ribociclib Plus Letrozole and, in Patients With a PIK3CA Mutation, on Second-line Treatment With Alpelisib Plus Fulvestrant (BioItaLEE)
Brief Title: Study of the Molecular Features of Postmenopausal Women With HR+ HER2-negative aBC on First-line Treatment With Ribociclib and Letrozole and, in Patients With a PIK3CA Mutation, on Second-line Treatment With Alpelisib Plus Fulvestrant
Acronym: BioItaLEE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011AIT01; 2017-004176-62 (EudraCT Number)
Record Dates: First submitted 2018-01-29; First posted 2018-02-20 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: HR-positive HER2-negative; advanced breast cancer; LEE011; ribociclib; letrozole; CDK; CDK4; CDK6; CDK4/6; Phase IIIb; ER-positive; PR-positive; postmenopausal; biomarker; ctDNA; liquid biopsy; PIK3CA; alpelisib; fulvestrant; BYL719
MeSH Terms: conditions — Breast Neoplasms; Hereditary Sensory and Autonomic Neuropathies | interventions — ribociclib; Letrozole; Alpelisib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ribociclib+letrozole (Experimental): Ribociclib oral (3weeks on/1week off) in combination with oral once daily letrozole: 600mg tablets ribociclib QD + 2.5 mg tablets letrozole QD
  Interventions: Drug: Ribociclib; Drug: Letrozole
- alpelisib+fulvestrant (Experimental): Alpelisib 300 mg oral daily on a continuous dosing schedule in combination with fulvestrant 500 mg intramuscular on Days 1 and 15 of Cycle 1, and on Day 1 of each cycle thereafter in a 28 days cycle
  Interventions: Drug: Alpelisib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Ribociclib — Ribociclib oral (3weeks on/1week off) in combination with oral once daily letrozole: 600mg tablets ribociclib QD + 2.5 mg tablets letrozole QD
  Other Names: LEE011
  Arms: ribociclib+letrozole
Drug: Letrozole — Ribociclib oral (3weeks on/1week off) in combination with oral once daily letrozole: 600mg tablets ribociclib QD + 2.5 mg tablets letrozole QD
  Arms: ribociclib+letrozole
Drug: Alpelisib — Alpelisib 300 mg oral daily on a continuous dosing schedule in combination with fulvestrant 500 mg intramuscular on Days 1 and 15 of Cycle 1, and on Day 1 of each cycle thereafter in a 28 days cycle
  Other Names: BYL719
  Arms: alpelisib+fulvestrant
Drug: Fulvestrant — Alpelisib 300 mg oral daily on a continuous dosing schedule in combination with fulvestrant 500 mg intramuscular on Days 1 and 15 of Cycle 1, and on Day 1 of each cycle thereafter in a 28 days cycle
  Arms: alpelisib+fulvestrant

SUMMARY:
The purpose of this clinical trial is to study of the molecular features of postmenopausal women with hormone receptor-positive (HR+) HER2-negative advanced breast cancer on first-line treatment with ribociclib and letrozole and, in patients with a PIK3CA mutation, on second-line treatment with alpelisib plus fulvestrant

DETAILED DESCRIPTION:
The main purpose of this local, multicenter study is to investigate genetic and gene expression alterations in tumor prior to and following progression on ribociclib, during core phase and then prior to and following progression on alpelisib and thus identify patterns of mutations, how they evolve, and their association with CDK4/6 inhibition and outcomes such as sustained response or early progression. The study also aims to evaluate pharmacogenomics and its association with adverse events (frequency and severity), drug-drug interactions and clinical outcomes.

Finally, the study will also generate additional long-term safety and efficacy data in this specific Italian population.

ELIGIBILITY:
CORE PHASE Inclusion Criteria:

* Patient has an advanced (locoregionally recurrent or metastatic) breast cancer in first line treatment (treatment naïve for the advanced setting).
* Patient is in post-menopause, defined by one of the following:
* Prior bilateral oophorectomy
* Age ≥60
* Age <60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifen, or ovarian suppression) and FSH and estradiol in the postmenopausal range per local normal range
* Patient has a histologically and/or cytologically confirmed diagnosis of estrogenreceptor positive and/or progesterone receptor positive breast cancer by local laboratory.
* Patient has an HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing.
* Patient is willing to undergo blood and tumor sample collection for the biological assessments/objectives as scheduled in the protocol.

CORE PHASE Exclusion Criteria:

* Patient who received prior treatment with any CDK4/6 inhibitor.
* Patient who received any prior systemic hormonal therapy or chemotherapy for advanced breast cancer.

Note:

Patients who received neo/adjuvant therapy for breast cancer are eligible. If the prior neo/adjuvant therapy included letrozole or anastrozole, the disease-free interval must be greater than 12 months from the completion of treatment until study entry.

• Patients who received ≤ 28 days of letrozole or anastrozole for advanced disease prior to inclusion in this trial are eligible.

- Patient is currently using other anti-cancer therapy. Other protocol-defined inclusion/exclusion criteria may apply.

EXTENSION PHASE Inclusion criteria:

* Patient has been discontinued (any reason allowed) from treatment with ribociclib + letrozole in the core phase and is deemed suitable for treatment with alpelisib + fulvestrant in second line. Ribociclib + letrozole must be the last treatment regimen before alpelisib + fulvestrant.
* Patient has PIK3CA mutation as determined in tumor tissue and/or plasma by a Novartis designated laboratory. Results of tissue samples obtained during the core phase (screening or EOT) are acceptable

EXTENSION PHASE Exclusion criteria:

* Patient has received prior treatment with any PI3K inhibitors.
* Patient is concurrently using other anti-cancer therapy. Ribociclib and letrozole used in the core phase must be discontinued at least 7 days prior to day one of the extension study treatment.

All drugs with overlapping toxicities must be discontinued within 7 days and AE resolved to NCI CTCAE v4.03 Grade ≤1 prior to study treatment. Exception to this criterion: patients with any grade of alopecia are allowed to enter the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 287 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline ctDNA alterations to progression disease during Core and Extension Phase | Up to approximately 36 months starting from Baseline of the core phase and Up to approximately 9 months starting from Baseline of the extension phase
  The percentage of patients with ctDNA alterations (i.e. such as but not limited to Rb, ESR1, cyclin D1, CDKN2A, PIK3CA, p53 and PTEN) will be provided over time to characterize the biological evolution of the disease in each patient. The association of these alterations with clinical outcomes will also be provided.

SECONDARY OUTCOMES:
Change from baseline serum TK1 concentrations to progression disease during core phase | Up to approximately 36 months starting from Baseline of the core phase
  Descriptive statistics of serum TK1 concentrations will be provided over time. The association/correlation of serum TK1 concentrations with clinical outcomes will also be provided.
The percentage of patients with ctDNA alterations will be provided over time in the subsets during Core and Extension Phase | Up to approximately 36 months starting from Baseline of the core phase and Up to approximately 9 months starting from Baseline of the extension phase
  The percentage of patients with ctDNA alterations will be provided over time in the subsets of long responder patients and those with early progression
Change from baseline tumor mutational burden (TMB) to progression disease during Core and Extension Phase | Up to approximately 36 months starting from Baseline of the core phase and Up to approximately 9 months starting from Baseline of the extension phase
  Descriptive statistics of tumor mutational burden (TMB), defined as a quantitative measure of the total number of ctDNA mutations per coding area of tumor genome, will be provided over time, according to the scheduled sample collections. The association of TMB values with clinical outcomes will also be provided.
The percentage of patients with mutations as assessed at baseline of the Core and Extension phase across different patient profiles | Screening Core Phase and Screening Extension Phase
  The percentage of patients with mutations as assessed at baseline by means of ctDNA sample, and tissue biopsy will be compared between the following patient profiles defined according to disease history (i.e. newly diagnosed vs. recurrent disease).
The percentage of patients with alterations detected through liquid biopsy vs. tissue biopsy during Core and Extension Phase | Up to approximately 36 months starting from Baseline of the core phase and Up to approximately 9 months starting from Baseline of the extension phase
  The percentage of patients with alterations detected at baseline and at disease progression will be compared between the two different procedures of detection (i.e. detection through liquid biopsy vs. tissue biopsy).
Change from baseline tumor microenvironment parameters to progression disease during Core and Extension Phase | Up to approximately 36 months starting from Baseline of the core phase and Up to approximately 9 months starting from Baseline of the extension phase
  Descriptive statistics of tumor microenvironment parameters on tumor biopsy will be provided at baseline and upon disease progression. The association of these tumor micro-environment parameters with clinical outcomes will also be provided.
Time-to-Progression (TTP) during Core and Extension Phase | Up to approximately 36 months starting from Baseline of the core phase and Up to approximately 9 months starting from Baseline of the extension phase
  Time to progression (TTP) is defined as time from date of start of treatment to the date of event defined as the first documented progression or death due to underlying cancer.
The number of patients with adverse events as a measure of safety and tolerability during Core and Extension Phase | Up to approximately 36 months starting from Baseline of the core phase and Up to approximately 9 months starting from Baseline of the extension phase
  Fequency and severity of AEs and SAEs
The percentage of patients with best overall response rate CR or PR during Core and Extension Phase | Up to approximately 36 months starting from Baseline of the core phase and Up to approximately 9 months starting from Baseline of the extension phase
  Overall response rate (ORR) is defined as the percentage of patients, with measurable disease, that showed best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1.
The percentage of patients with clinical benefit during Core and Extension Phase | Up to approximately 36 months starting from Baseline of the core phase and Up to approximately 9 months starting from Baseline of the extension phase
  Clinical benefit rate (CBR) is defined as the percentage of patients with a best overall response of complete response (CR), or partial response (PR) or an overall lesion response of stable disease (SD), lasting as per local review, for a duration of at least 24 weeks. CR, PR and SD are defined according to RECIST 1.1.
The percentage of participants with adverse events as a measure of safety and tolerability during Core and Extension Phase | Up to approximately 36 months starting from Baseline of the core phase and Up to approximately 9 months starting from Baseline of the extension phase
  Frequency and severity of AEs and SAEs

CONTACTS AND LOCATIONS:
Locations (34):
- Italy (34):
  - Novartis Investigative Site, Casale Monferrato, AL
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Benevento, BN
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brindisi, BR
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, San Giovanni Rotondo, FG
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Livorno, LI
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Macerata, MC
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Nuoro, NU
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Prato, PO
  - Novartis Investigative Site, Fano, PU
  - Novartis Investigative Site, Faenza, RA
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Candiolo, TO
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Negrar, VR
  - Novartis Investigative Site, Napoli

IPD SHARING:
Plan to Share IPD: Undecided